CLINICAL TRIAL: NCT07053371
Title: Effectiveness of Peanut Ball During the First Stage of Labor on Maternal and Neonatal Outcomes
Brief Title: Peanut Ball During the First Stage of Labor
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Peanut Ball during labor Stage
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Labor Duration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Women in this group to utilize peanut birth balls
  Interventions: Other: Peanut birth ball
- Control group (No Intervention): The control group received conventional hospital care from their obstetrician.

INTERVENTIONS:
Other: Peanut birth ball — The 45 x 80 cm peanut birth ball was positioned between the woman's legs during the first stage's active phase, starting at 4 cm cervical dilatation for the intervention group
  Arms: Intervention group

SUMMARY:
The current study aimed to assess the effectiveness of peanut ball during first stage of labor on maternal and neonatal outcomes.

DETAILED DESCRIPTION:
Labor, the climax of pregnancy, involves specialized care that covers women's social, physiological, anatomical, and emotional demands. Comfort must always come first throughout labor, and supportive techniques are essential from the prodromal to the expulsive phases.

The painful uterine contractions that precede the entire cervical dilatation characterize the 1st stage of labor. The 1st stage of labor consists of three stages: the latent phase, the active phase, and the transition period. The uterine tissues' distension and the cervix's dilatation are the causes of the cramp-like contraction discomfort at this stage, which is transmitted to the abdomen and lumbosacral regions by spinal nerves.

Stress brought on by labor pain might result in an excess of stress chemicals like catecholamines and steroids. This hormone can increase blood vessel vasoconstriction and smooth muscle tension, which can halt uterine contractions, lower uteroplacental circulation, and reduce the uterus's blood supply and oxygen, all of which exacerbate pain perceptions. The blood concentration of catecholamines rises with prolonged delivery.

The appropriate management of labor pain continues to be one of the most important aspects of intrapartum care. Therefore, enhancing the comfort of mothers giving birth is one of the most important responsibilities of nurses and other healthcare professionals. Women might feel comfort and control during childbirth if health issues are less common. Many efforts have been made to improve the outcomes of mother and newborn births and to reduce the duration of labor.

Changes in posture and freedom of mobility are useful strategies to lessen the impact of labor pain. During the prenatal period, posture changes and techniques to control labor pain should be taught. Pregnant women who were not educated throughout the prenatal period should be informed about the importance of movement and position changes during the latent phase of labor and when pain is at its lowest and communication is at its highest.

Numerous physiological measures were implemented to shorten the length of labor including pelvic rocking, deep breathing exercises, pregnancy exercises, and birthing ball exercises. Frequent position adjustments and movements during labor are recommended by the World Health Organization (WHO) as a way to reduce prolonged labor and avoid cesarean sections. To address these issues and put WHO recommendations into practice, the peanut birth ball could be a useful tool for routine position modifications without interfering with labor procedures.

Peanut balls are presented as a new strategy for improving women's labor and delivery outcomes. Although women have used birthing balls to advance labor for many years, the peanut ball is available in different sizes to make sure that women will find it comfortable. Furthermore, for women who have had an epidural, the peanut ball may be utilized in four different postures depending on the fetal station and stage of labor. Furthermore, it has the advantages of being affordable, reusable, and noninvasive.

Because the elasticity of the ball stimulates endorphin receptors in the pelvis, sitting and swinging on it makes the woman feel more at ease and encourages the release of endorphins. Additionally, the expansion and relaxation of pelvic muscles and bones, as well as the process of delivery, are aided by gravity, which improves fetal descent.

Maternity nurses play a crucial role in ensuring safe and normal childbirth. They need to closely monitor the progress of labor to facilitate a smooth delivery. Furthermore, satisfying the woman's emotional requirements following her physical demands will enable a happy delivery experience and contribute to the safe commencement of mother-infant bonding..

ELIGIBILITY:
Inclusion Criteria:

* Low-risk primipara in active phase of labor, aged 20 -35 years with single living fetus in cephalic presentation and full-term pregnancy which lasts between 37-42 weeks

Exclusion Criteria:

* Women with medical or obstetric complications were excluded from the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Parturient women
Enrollment: 104 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progress of labor, duration of each stage | During the active phase of labor
  Analysis of the progress of labor and the duration of labor stages

REFERENCES:
- [Background] Hickey L, Savage J. Effect of Peanut Ball and Position Changes in Women Laboring With an Epidural. Nurs Womens Health. 2019 Jun;23(3):245-252. doi: 10.1016/j.nwh.2019.04.004. Epub 2019 May 9. PMID 31077640
- [Background] Mercier RJ, Kwan M. Impact of Peanut Ball Device on the Duration of Active Labor: A Randomized Control Trial. Am J Perinatol. 2018 Aug;35(10):1006-1011. doi: 10.1055/s-0038-1636531. Epub 2018 Mar 6. PMID 29510425
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29510425/